CLINICAL TRIAL: NCT06841666
Title: Evaluating the Efficacy of Atomoxetine in Reducing Primary Nocturnal Enuresis in Children With ADHD
Brief Title: Evaluating the Efficacy of Atomoxetine in Reducing Primary Nocturnal Enuresis in Children With ADHD: A Randomized, Placebo-Controlled Study
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Ibrahim Younes, lecturer of psychiatry, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 36264؛ٌ1054/1/25
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: ADHD; Primary Nocturnal Enuresis
Keywords: Primary Nocturnal Enuresis; ADHD; Atomoxetine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: A Randomized, Placebo-Controlled Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Treatment) (Experimental): 50 patients will recieve Atomoxetine, 0.5-1.2 mg/kg/day, administered in the evening for six months.
  Frequency of nocturnal enuresis episodes, recorded by parents in a nightly log. ADHD symptoms, assessed using Conners-48 scores at baseline, 1, 3, and 6 months.
  Interventions: Drug: Atomoxetine
- Group 2 (Control) (Experimental): 50 participants will receive Placebo identical in form and dosing schedule. for 6 months.
  Frequency of nocturnal enuresis episodes, recorded by parents in a nightly log. ADHD symptoms, assessed using Conners-48 scores at baseline, 1, 3, and 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Atomoxetine, 0.5-1.2 mg/kg/day, administered in the evening for six months.
  Arms: Group 1 (Treatment)
Drug: Placebo — Placebo identical in form and dosing schedule for six months.
  Arms: Group 2 (Control)

SUMMARY:
1. Primary Aim: To evaluate the efficacy of atomoxetine in reducing the frequency of primary nocturnal enuresis episodes in children with ADHD.
2. Secondary Aim: To determine if improvements in attention symptoms correlate with reductions in nocturnal enuresis episodes.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a prevalent neurodevelopmental disorder affecting approximately 5-7% of school-aged children globally. It is characterized by inattention, hyperactivity, and impulsivity, impairing academic, social, and daily functioning (American Psychiatric Association, 2013). The Conners-48 scale is frequently used to assess ADHD severity, offering a standardized tool for research and clinical practice. Treatments for ADHD often combine behavioral therapies with pharmacological agents such as stimulants or non-stimulants, including atomoxetine (Cortese et al., 2016).

Primary nocturnal enuresis (PNE) refers to involuntary urination during sleep in children aged five or older, without any underlying organic or neurological disorder. While PNE typically diminishes with age, its persistence can cause significant psychosocial stress for children and their families. Studies suggest that children with ADHD experience PNE at higher rates than their neurotypical peers, underscoring the need for tailored management strategies (Hagerty et al., 2015).

Interrelationship Between ADHD and Enuresis:

Shared neurobiological pathways may explain the coexistence of ADHD and PNE. Both conditions involve dysregulation in arousal and inhibitory control mechanisms, leading to disrupted sleep patterns and impaired bladder control during sleep (Shreeram et al., 2009). Despite this overlap, current treatment paradigms rarely address both conditions concurrently, leaving a clinical gap in care.

Rationale for Atomoxetine in PNE:

Atomoxetine, a selective norepinephrine reuptake inhibitor, is a non-stimulant ADHD medication effective for managing attention deficits and impulsivity. It may also influence bladder control by enhancing norepinephrine activity in brainstem regions implicated in micturition (Kim et al., 2015). This potential dual benefit positions atomoxetine as a promising treatment option for ADHD and comorbid PNE.

Clinical and Research Gap:

Although extensive research has validated atomoxetine's efficacy for ADHD, limited studies explore its effects on comorbid conditions like PNE. This study aims to evaluate the frequency of nocturnal enuresis episodes and changes in ADHD symptoms, providing insight into atomoxetine's potential dual benefits. Findings may inform integrated therapeutic approaches for children with ADHD and PNE.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years diagnosed with ADHD per Conners-48 scale. Children experiencing primary nocturnal enuresis.

Exclusion Criteria:

* Secondary causes of enuresis (e.g., urinary tract infections, diabetes). Use of other enuresis treatments. Known contraindications to atomoxetine.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of nocturnal enuresis episodes, recorded by parents in a nightly log. | 6months
  * Baseline data: enuresis frequency.
  * Follow-up assessments at 1, 3, and 6 months:
  Parent-maintained logs of enuresis episodes.

SECONDARY OUTCOMES:
ADHD symptoms, assessed using Conners-48 scores at baseline, 1, 3, and 6 months | 6months
  * Baseline data: demographic details, ADHD severity (Conners-48),
  * Follow-up assessments at 1, 3, and 6 months:
    * Conners-48 scores to monitor ADHD symptom changes.

REFERENCES:
- [Result] Meredith SE, Juliano LM, Hughes JR, Griffiths RR. Caffeine Use Disorder: A Comprehensive Review and Research Agenda. J Caffeine Res. 2013 Sep;3(3):114-130. doi: 10.1089/jcr.2013.0016. PMID 24761279